CLINICAL TRIAL: NCT04616222
Title: A Retrospective Comparison of the Efficacy and Safety of Celsior® in Pediatric Cardiac Surgery for Transposition of the Great Vessels
Acronym: CELSIOR-TGV
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: CELSIOR-TGV_2020
Record Dates: First submitted 2020-07-23; First posted 2020-11-04 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-07

CONDITIONS: Transposition of Great Vessels
MeSH Terms: conditions — Transposition of Great Vessels

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CELSIOR® group: Patient who received Celsior® during their transposition of the great vessels surgery
  Interventions: Drug: CELSIOR® group
- Saint-Thomas group: Patient who received Saint-Thomas during their transposition of the great vessels surgery
  Interventions: Drug: Saint-Thomas group

INTERVENTIONS:
Drug: CELSIOR® group — Patient who received Celsior® during their transposition of the great vessels surgery according to the routine care.
  Groups: CELSIOR® group
Drug: Saint-Thomas group — Patient who received Saint-Thomas during their transposition of the great vessels surgery according to the routine care.
  Groups: Saint-Thomas group

SUMMARY:
Celsior® is an organ preservation solution used for the harvesting and the preservation of solid organs. Its use as a crystalloid cardioplegia solution has been established recently. Its main advantage is the long duration of myocardial protection. Compared to the other cardioplegia solutions, it allows a reduced amount of solution administered during the surgery and fewer interruptions during the intervention for the administration of supplemental doses of cardioplegia for long and complex operations.

The objective of this register is to compare the safety and the efficacy of Celsior® to the old cardioplegia solution Saint-Thomas used as cardioplegia solution in surgery of the transposition of great vessels, the arterial switch operation.

ELIGIBILITY:
Inclusion Criteria:

* Patient of neonatal age at the time of the intervention
* Patients with a transposition of the great vessels with intact septum and with the arterial switch operation performed as a corrective procedure
* CELSIOR® used as cardioplegia solution between 2012 and 2019
* Saint-Thomas used as cardioplegia solution (control group) between 2005 and 2011

Exclusion Criteria:

* Major cardiovascular malformations needing correction during the surgery for the transposition of great vessels including : interventricular communication, coarctation of the aorta, interruption of the aortic arch
* Significant anomalies of coronary arteries origin or paths including : intramural course, single coronary ostium
* Opposition to participate in this retrospective research

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Paediatric patients with an arterial switch operation for transposition of the great vessels
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2020-12-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Death at 30 days after surgery | 30 days
  Death at 30 days after surgery

SECONDARY OUTCOMES:
Post-operative troponin levels | 48 hours
  Troponin in ng/L
Cardiac rhythm assessment | 24 hours
  Percentage of abnormal rhythm
Variation of pre- and post-operative creatinine levels | 24 hours
  Creatinine in µmol/L
Intensive care unit length of stay | 30 days
  In days

CONTACTS AND LOCATIONS:
Locations (1):
- : Hôpital Louis Pradel - Service de Chirurgie Cardiaque C, Bron, France

REFERENCES:
- [Derived] Bulescu NC, Mitchell J, Metton O, El Jonhy N, Amaz C, Perouse de Montclos T, Lilot M, Mewton N, Henaine R. Celsior(R) vs. St Thomas(R) cardioplegia: analysis of myocardial protection and clinical safety in neonates. Front Pediatr. 2024 Jul 8;12:1430832. doi: 10.3389/fped.2024.1430832. eCollection 2024. PMID 39040670